CLINICAL TRIAL: NCT01351324
Title: Acute Elevation of Non-esterified Fatty Acids on Endothelial Function and Insulin Sensitivity: A Comparison of Saturated and Long Chain n-3 Polyunsaturated Fatty Acids During the Postprandial Phase
Brief Title: A Study of Different Types of Fatty Acid on Risk Factors for Heart Disease
Acronym: eFAIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Unilever R&D (Industry); Foundation for Research Science and Technology (New Zealand) (Unknown)
Responsible Party: Professor Christine Williams, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CMW-BB/E021816/1
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-04

CONDITIONS: Cardiovascular Risk Factors
Keywords: Endothelial function; Non-esterified fatty acids; Insulin sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SFA (Experimental): Oral dose of palmitic acid (SFA) given as a chocolate-flavoured drink every 30 min (0-390 min) with a continuous infusion of heparin (60-390 min).
  Interventions: Dietary Supplement: Absence or presence of fish oil
- SFA + LC n-3 PUFA (Experimental): Oral dose of palmitic acid and DHA-rich fish oil (SFA + LC n-3 PUFA) given as a chocolate-flavoured drink every 30 min (0-390 min) together with a continuous infusion of heparin (60-390 min).
  Interventions: Dietary Supplement: Absence or presence of fish oil

INTERVENTIONS:
Dietary Supplement: Absence or presence of fish oil — Oral dose of saturated fat with or without fish oil and a heparin infusion

SUMMARY:
Experimental elevation of non-esterified fatty acids (NEFA) impairs endothelial function and insulin sensitivity but the impact of NEFA composition is unknown.

The objective was to test the effect of acute elevation of NEFA enriched with either saturated fatty acids (SFA) or SFA with long-chain n-3 polyunsaturated fatty acids (LC n-3 PUFA) on postprandial vascular function measured via flow-mediated dilatation (FMD), laser Doppler iontophoresis (LDI) and digital volume pulse (DVP), followed by a hyperinsulinaemic-euglycaemic clamp as a measure of whole body insulin sensitivity.

DETAILED DESCRIPTION:
To investigate potential diet-gene interactions, potential subjects (n=370) were prospectively genotyped for the eNOS Glu298Asp polymorphism, of which 35 were Asp298 and 150 were Glu298 homozygotes. Three subjects in the Asp298 group were unable to participate, two were unsuitable according to selection criteria and one subject subsequently withdrew from the study. Subjects homozygous for Asp298 (n=29) and Glu298 (n=30) were therefore selected, balanced for gender, age and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Either homozygous for eNOS Glu298 (wildtype)or eNOS Asp298 (variant)

Exclusion Criteria:

* Smokers
* Raised fasting blood lipids
* Taking excessive fish oil supplements (>1g EPA/DHA per day)
* Taking medication known to influence blood lipids, blood pressure or blood clotting

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilatation | Change from baseline to 240 min
Flow-mediated dilatation | Change from 240 min to 390 min

SECONDARY OUTCOMES:
Digital volume pulse | Change from baseline to 240 min
Laser Doppler iontophoresis | Change from baseline to 240 min
Insulin sensitivity | 390 min
NEFA composition | Change from baseline to 240 min
Circulating endothelial function markers | Change from baseline to 240 min
Digital volume pulse | Change from 240 min to 390 min
Laser Doppler iontophoresis | Change from 240 min to 390 min
Circulating endothelial markers | Change from 240 min to 390 min

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Williams, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

REFERENCES:
- [Derived] Newens KJ, Thompson AK, Jackson KG, Williams CM. Endothelial function and insulin sensitivity during acute non-esterified fatty acid elevation: Effects of fat composition and gender. Nutr Metab Cardiovasc Dis. 2015 Jun;25(6):575-81. doi: 10.1016/j.numecd.2015.03.004. Epub 2015 Mar 14. PMID 25921849
- [Derived] Newens KJ, Thompson AK, Jackson KG, Wright J, Williams CM. DHA-rich fish oil reverses the detrimental effects of saturated fatty acids on postprandial vascular reactivity. Am J Clin Nutr. 2011 Sep;94(3):742-8. doi: 10.3945/ajcn.110.009233. Epub 2011 Aug 10. PMID 21831993